CLINICAL TRIAL: NCT03604731
Title: Persistent Multiorgan Failure in Intensive Care Units: Risk Factors, Prognosis, Outcomes
Brief Title: Persistent Multiorgan Failure in Intensive Care Units
Acronym: PROPOSe
Status: Completed | Type: Observational
Sponsor: Research Institute for Complex Problems of Cardiovascular Diseases, Russia (Other)
Responsible Party: Principal Investigator, Evgeny Grigoryev, clinical professor, Research Institute for Complex Problems of Cardiovascular Diseases, Russia
Other Study IDs: 201721
Record Dates: First submitted 2018-07-19; First posted 2018-07-27 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Systemic Inflammatory Response Syndrome; Sepsis; Multiorgan Failure
Keywords: Immunology, Suppression, Inflammation, Cardiac, Surgery
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Sepsis; Multiple Organ Failure; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Blood serum (cytokines, mit DNA)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Uncomplicated cardiac surgery patients: Patients after schedulled cardiac surgery procedures
- Complicated cardiac surgery patients: Patients after schedulled cardiac surgery procedures complicated by multiorgan failure
  Interventions: Device: cytokine adsorbtion during extracorporeal circulation

INTERVENTIONS:
Device: cytokine adsorbtion during extracorporeal circulation — preventive use of cytokine adsorption and modulation of the cytokine response in the course of artificial circulation
  Groups: Complicated cardiac surgery patients

SUMMARY:
Multiorgan failure (MOF) as a result of any critical condition is a complex set of immunological and biochemical interactions leading to death in patients who are effectively subjected to primary resuscitation (correction of circulatory hypoxia in trauma and blood loss, restoration of blood circulation after operations with artificial circulation. The frequency of MOF varies depending on the primary diagnosis of a critical patient and, according to a number of authors, is 60% for sepsis, and for severe co-occurring trauma up to 40% of all critical patients. However, if one remembers that the MOF is verified only by clinical scales of assessing the severity of the patient's condition, which presupposes the presence of the already existing pathophysiological mechanisms of MOF as multi-organ dysfunction, it is possible to declare a 100% presence of MOF in all critical patients. The data of Graetz et al (2016) show that none of the available three variants of pathophysiological mechanisms (anomaly of microcirculation, persistent inflammation, immune suppression and catabolism, cellular hibernation and staning) have been unambiguously demonstrated, which also reflected the lack of effectiveness of methods therapy, proposed, based on the pathogenesis options for MOF. A so-called danger-model has a special place in the genesis of the persistence of the MOF, which justifies an active search for distress-associated and pathogen-associated molecular patterns for their objectification and probable elimination. The systemic inflammatory response in patients. included in the study, is not a primary infection. It is also important to determine the role of danger-associated molecular patterns (DAMP) in the genesis of immune suppression as the leading immunological phenotype of MOF in later periods and to evaluate the relationship between DAMP expression and immunosuppressive cells of monocyte origin. The study has a mixed (retro- and prospective) character.

DETAILED DESCRIPTION:
1. Based on the patient database analysis, by the method of continuous sampling of the cardiac surgery patients to the intensive care unit for the period 2006-2018, to determine the clinical risk factors for the development of a persistent MOF (MOF + persistent MOF, which lasts more than 7 days and is determined primarily by based on indicators of objective assessment of the patient's condition - the SOFA scale is more than 8 points on the 7th day of the critical care). To form a prognostic model.
2. By means of biochemical analysis of blood serum and cells, identify biological markers MES specific for distant organs and supplement the prognostic model of persistent MOF. It is planned to detect serum concentrations (1) of surfactant protein A (organ-specific lung marker for the development of acute respiratory distress syndrome as manifestations of MOF), (2) intestinal fatty acid binding protein (organ-specific marker of acute intestinal distress (3) S100 protein - a marker of brain damage) with an assessment of prognostic and diagnostic significance with respect to the MOF.
3. To assess the prognostic and diagnostic significance of serum mitochondrial DNA as one of the variants of the danger-associated molecular pattern.
4. To characterize the presence of an immunosuppressive phenotype of a critical patient with MOF by examining the expression and serum concentration of: (a) myeloid suppressor cells; (b) T-reg cells expressing CD39; (c) CD62 and CD11b expression on neutrophils on monocytes; (d) soluble sTREM-1, (e) HLA-DR on monocytes. In addition, it will be planned to study the "classic" serum cytokines (tumor necrosis factor alpha, interleukin 1,6,8,10, HMGB-1).
5. On the basis of the diagnostic panel obtained, to try to conduct an individualized choice of methods of preventive therapy for MOF. It is proposed to use: (1) cytokine modulation of the systemic inflammatory response by sorption of cytokines on selective sorbents, (2) cytokine modulation by sorption of cytokines on polymethylmethacrylate membranes. It is assumed that in order for these methods to be preventative, they should be used not only in conditions of treatment in the intensive care unit, but also in the operating room at the time of extracorporeal perfusion.

ELIGIBILITY:
Inclusion Criteria:

* patients after planned cardiac surgey
* informed consent

Exclusion Criteria:

* age less 18 and more then 80 years
* unplanned cardiac surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated on the heart and trunk vessels under conditions of artificial circulation (coronary artery bypass grafting, prosthetic / cardiac valve repair, operations on the aorta and its branches)
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Intensive Care Unit (ICU) 28 day mortality | 28 day
  Mortality in ICU period within 28 day

SECONDARY OUTCOMES:
Free of multiorgan failure (MOF) days | 28 day
  Free of MOF period within 28 day
Mechanical ventilation (MV) - dependent days | 28 day
  MV dependens period within 28 day
Renal Replacement Therapy (RRT) dependens | 28 day
  Renal Replacement Therapy period within 28 day
Assosiation of severity of ilness | 28 day
  Sequential Organ Failure Assesment

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hotchkiss RS, Moldawer LL, Opal SM, Reinhart K, Turnbull IR, Vincent JL. Sepsis and septic shock. Nat Rev Dis Primers. 2016 Jun 30;2:16045. doi: 10.1038/nrdp.2016.45. PMID 28117397
- [Background] Gaudilliere B, Angst MS, Hotchkiss RS. Deep Immune Profiling in Trauma and Sepsis: Flow Is the Way to Go! Crit Care Med. 2017 Sep;45(9):1577-1578. doi: 10.1097/CCM.0000000000002594. No abstract available. PMID 28816846
- [Background] Graetz TJ, Hotchkiss RS. Sepsis: Preventing organ failure in sepsis - the search continues. Nat Rev Nephrol. 2017 Jan;13(1):5-6. doi: 10.1038/nrneph.2016.171. Epub 2016 Nov 21. PMID 27867191
- [Background] Asehnoune K, Hotchkiss RS, Monneret G. Understanding why clinicians should care about danger-associated molecular patterns. Intensive Care Med. 2016 Apr;42(4):611-614. doi: 10.1007/s00134-015-4198-y. Epub 2016 Feb 24. No abstract available. PMID 26912314
- [Background] Malard B, Lambert C, Kellum JA. In vitro comparison of the adsorption of inflammatory mediators by blood purification devices. Intensive Care Med Exp. 2018 May 4;6(1):12. doi: 10.1186/s40635-018-0177-2. PMID 29728790
- [Background] Rosenthal M, Gabrielli A, Moore F. The evolution of nutritional support in long term ICU patients: from multisystem organ failure to persistent inflammation immunosuppression catabolism syndrome. Minerva Anestesiol. 2016 Jan;82(1):84-96. Epub 2015 Feb 20. PMID 25697882